CLINICAL TRIAL: NCT03606590
Title: HEPANOVA: a Phase II Trial of Tumor Treating Fields (TTFields, 150kHz) Concomitant with Sorafenib for Advanced Hepatocellular Carcinoma (HCC)
Brief Title: Effect of Tumor Treating Fields (TTFields, 150kHz) Concomitant with Sorafenib for Advanced Hepatocellular Carcinoma (HCC) (HEPANOVA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NovoCure Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EF-30
Record Dates: First submitted 2018-07-23; First posted 2018-07-31 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Treatment; Minimal toxicity; TTFields; Tumor Treating Fields; Novocure; Sorafenib; Nexavar
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TTFields in combination with sorafenib (Experimental): Patients will be treated continuously with TTFields, in addition to sorafenib
  Interventions: Device: NovoTTF-100L(P) device; Drug: Sorafenib

INTERVENTIONS:
Device: NovoTTF-100L(P) device — Patients will be treated continuously with the NovoTTF-100L(P) device. NovoTTF-100L(P) treatment will consist of wearing four electrically insulated electrode arrays on the abdomen. The treatment enables the patient to maintain regular daily routine.
  Other Names: TTFields
Drug: Sorafenib — Sorafenib 400 mg (2 x 200 mg tablets) taken twice daily without food (at least 1 hour before or 2 hours after a meal).
  Other Names: Nexavar

SUMMARY:
The study is a prospective, phase II trial single arm, historical control aimed to test the efficacy and safety of TTFields, using the NovoTTF-100L(P) System, in combination with sorafenib in patient with advanced HCC. The device is an experimental, portable, battery operated device for chronic administration of alternating electric fields (termed TTFields or TTF) to the region of the malignant tumor, by means of surface, insulated electrode arrays.

DETAILED DESCRIPTION:
PAST PRE-CLINICAL AND CLINICAL EXPERIENCE:

The effect of the electric fields (TTFields, TTF) has demonstrated significant activity in in vitro hepatocellular carcinoma pre-clinical models. In addition, TTFields have shown to inhibit metastatic spread of malignant melanoma in in vivo experiment.

In pilot study, 40 patients with locally advanced or metastatic pancreatic adenocarcinoma received chemotherapy with TTFields (150 kHz) applied to the abdomen. The combination was well tolerated and the only device-related adverse event was contact dermatitis.

In addition, a phase III trial of Optune® (200 kHz) as monotherapy compared to active chemotherapy in recurrent glioblastoma patients showed TTFields to be equivalent to active chemotherapy in extending survival, associated with minimal toxicity, good quality of life, and activity within the brain (14% response rate) (Stupp R., et al., EJC 2012). Finally, a phase III trial of Optune® combined with maintenance temozolomide compared to maintenance temozolomide alone has shown that combined therapy led to a significant improvement in both progression free survival and overall survival in patients with newly diagnosed glioblastoma without the addition of high grade toxicity and without decline in quality of life (Stupp R., et al., JAMA 2017).

DESCRIPTION OF THE TRIAL:

All patients included in this trial are patients with locally advanced hepatocellular carcinoma. In addition, all patients must meet all eligibility criteria.

Eligible patients will be enrolled, baseline tests will be performed and the patients will be treated continuously with the device concomitant with sorafenib until disease progression in the liver.

TTFields treatment will consist of wearing four electrically insulated electrode arrays on the abdomen. Electrode array placement will require shaving of the abdomen/back as necessary before and during the treatment. After an initial short visit to the clinic for training and monitoring, patients will be released to continue treatment at home where they can maintain their regular daily routine.

During the trial the patient will need to return once every 4 weeks to the clinic where an examination by a physician and a routine laboratory examinations will be done. These routine visits will continue for as long as the patient's disease is not progressing in the liver. A routine CT or MRI scan of the abdomen will be performed at baseline and every 12 weeks thereafter, until disease progression in the liver. After this follow up plan, patients will be contacted once per month by telephone to answer basic questions about their health status.

SCIENTIFIC BACKGROUND:

Electric fields exert forces on electric charges similar to the way a magnet exerts forces on metallic particles within a magnetic field. These forces cause movement and rotation of electrically charged biological building blocks, much like the alignment of metallic particles seen along the lines of force radiating outwards from a magnet.

Electric fields can also cause muscles to twitch and if strong enough may heat tissues. TTFields are alternating electric fields of low intensity. This means that they change their direction repetitively many times a second. Since they change direction very rapidly (150 thousand times a second), they do not cause muscles to twitch, nor do they have any effects on other electrically activated tissues in the body (brain, nerves and heart). Since the intensities of TTFields in the body are very low, they do not cause heating.

The breakthrough finding made by Novocure was that finely tuned alternating fields of very low intensity, now termed TTFields (Tumor Treating Fields), cause a significant slowing in the growth of cancer cells. Due to the unique geometric shape of cancer cells when they are multiplying, TTFields cause electrically-charged cellular components of these cells to change their location within the dividing cell, disrupting their normal function and ultimately leading to cell death. In addition, cancer cells also contain miniature building blocks which act as tiny motors in moving essential parts of the cells from place to place. TTFields interfere with the normal orientation of these tiny motors related to other cellular components since they are electrically-charged as well. As a result of these two effects, tumor cell division is slowed, results in cellular death or reverses after continuous exposure to TTFields.

Other cells in the body (normal healthy tissues) are affected much less than cancer cells since they multiply at a much slower rate if at all. In addition TTFields can be directed to a certain part of the body, leaving sensitive areas out of their reach. Finally, the frequency of TTFields applied to each type of cancer is specific and may not damage normally dividing cells in healthy tissues.

In conclusion, TTFields hold the promise of serving as a brand new treatment for hepatocellular carcinoma with very few side effects.

ELIGIBILITY:
Inclusion Criteria:

1. HCC diagnosed by biopsy, or by imaging criteria (CT/MRI) and AFP
2. ≥ 18 years of age
3. Barcelona Clinic Liver Cancer Staging (BCLC) Stage 0-C
4. Child-Turcotte-Pugh (CTP) score between 5 and 8 points
5. Measurable disease per RECIST Criteria
6. At least 4 weeks since major surgery
7. ECOG Performance Status (PS) of 0-2
8. Life expectancy of at least 12 weeks
9. All subjects must sign written informed consent
10. Able to operate the NovoTTF-100L(P) System independently or with the help of a caregiver.

Exclusion Criteria:

1. Patient candidate for surgical resection or local treatment (e.g. TACE, SIRT, RFTA, microwave, surgery)
2. High levels of serum HBV DNA without anti-viral therapy
3. Prior malignancy requiring anti-tumor treatment (apart from in-situ cervical cancer, in situ breast cancer, non-melanomatous skin cancers, or any malignancy for which treatment was received and there is no evidence of disease for at least 5 years) or concurrent malignancy.
4. Significant co-morbidities within 4 weeks prior to enrollment, including the following:

   1. neurologic or psychiatric disorders such as dementia and uncontrolled seizures
   2. active, uncontrolled infections
   3. active, disseminated coagulation disorder
   4. Significant renal impairment
   5. Clinically significant cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia)
   6. Chronic diarrhea
   7. History of any psychological or psychiatric condition that might impair the patient's ability to understand or comply with the requirements of the study or to provide consent.
   8. Other co-morbidities deemed by the investigator as such that may impact the compliance of the patient with the study protocol and follow up
5. Implanted pacemaker, defibrillator or other electrical medical devices in the torso
6. Known allergies to medical adhesives or hydrogel
7. Pregnant or breast feeding (all patients of childbearing potential must use effective contraception method during the entire period of the study based on the recommendation of the investigator or a gynecologist)
8. Admitted to an institution by administrative or court order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2021-01-14 (Actual)

PRIMARY OUTCOMES:
Overall response rate | 30 months
  The percentage of patients who had either complete response or partial response per RECIST criteria following enrollment in the trial.

SECONDARY OUTCOMES:
In-field control rate at one year | 12 months
  The percentage of patients who did not have progression confined to the right hypochondriac and epigastric anatomical regions (defined by the diaphragm as a superior border, the left midclavicular line as a lateral border and the subcostal plane as an inferior border) per RECIST criteria at one year following the time of enrollment in the trial, or death.
Overall survival | 30 months
  The time from enrollment in the trial until date of death.
Progression Free Survival | 30 months
  The time from enrollment in the trial until progression per RECIST Criteria or death.
Distant metastases-free survival rate at 1 year | 12 months
  The percentage of patients who did not have new metastases outside of the liver (compared to the baseline CT/MRI) at one year following the time of enrollment in the trial, or death.
Overall survival at one year | 12 months
  The percentage of patients who are alive at one year following the time of enrollment in the trial.
Progression free survival at 6 and 12 months | 12 months
  the percentage of patients who are not progressive per RECIST Criteria, or dead at 6 and 12 months following the time of enrollment in the trial.
Severity and frequency of adverse events | 30 months
  Incidence of adverse event out of the number of patients who receive at least 1 day of TTFields treatment.

CONTACTS AND LOCATIONS:
Locations (8):
- University Hospital Fakultni Nemocnice Olomouc, Oncology Clinic, Olomouc, Czechia
- CHU de Nantes, Nantes, France
- Germany (2):
  - University Medical Center - University of Freiburg, Freiburg im Breisgau
  - Ulm University Hospital, Ulm
- Università Campus Bio-Medico di Roma, Rome, Italy
- Uniwersytet Medyczny im. Karola Marcinkowskiego w Poznaniu, Poznan, Poland
- Spain (2):
  - Vall d'Hebron Institute of Oncology (VHIO), Barcelona
  - HM Hospitales - Centro Integral Oncológico Clara Campal, Madrid

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kirson ED, Gurvich Z, Schneiderman R, Dekel E, Itzhaki A, Wasserman Y, Schatzberger R, Palti Y. Disruption of cancer cell replication by alternating electric fields. Cancer Res. 2004 May 1;64(9):3288-95. doi: 10.1158/0008-5472.can-04-0083. PMID 15126372
- [Background] Kirson ED, Dbaly V, Tovarys F, Vymazal J, Soustiel JF, Itzhaki A, Mordechovich D, Steinberg-Shapira S, Gurvich Z, Schneiderman R, Wasserman Y, Salzberg M, Ryffel B, Goldsher D, Dekel E, Palti Y. Alternating electric fields arrest cell proliferation in animal tumor models and human brain tumors. Proc Natl Acad Sci U S A. 2007 Jun 12;104(24):10152-7. doi: 10.1073/pnas.0702916104. Epub 2007 Jun 5. PMID 17551011
- [Background] Stupp R, Wong ET, Kanner AA, Steinberg D, Engelhard H, Heidecke V, Kirson ED, Taillibert S, Liebermann F, Dbaly V, Ram Z, Villano JL, Rainov N, Weinberg U, Schiff D, Kunschner L, Raizer J, Honnorat J, Sloan A, Malkin M, Landolfi JC, Payer F, Mehdorn M, Weil RJ, Pannullo SC, Westphal M, Smrcka M, Chin L, Kostron H, Hofer S, Bruce J, Cosgrove R, Paleologous N, Palti Y, Gutin PH. NovoTTF-100A versus physician's choice chemotherapy in recurrent glioblastoma: a randomised phase III trial of a novel treatment modality. Eur J Cancer. 2012 Sep;48(14):2192-202. doi: 10.1016/j.ejca.2012.04.011. Epub 2012 May 18. PMID 22608262
- [Background] Kirson ED, Giladi M, Gurvich Z, Itzhaki A, Mordechovich D, Schneiderman RS, Wasserman Y, Ryffel B, Goldsher D, Palti Y. Alternating electric fields (TTFields) inhibit metastatic spread of solid tumors to the lungs. Clin Exp Metastasis. 2009;26(7):633-40. doi: 10.1007/s10585-009-9262-y. Epub 2009 Apr 23. PMID 19387848
- [Background] Giladi M, Schneiderman RS, Voloshin T, Porat Y, Munster M, Blat R, Sherbo S, Bomzon Z, Urman N, Itzhaki A, Cahal S, Shteingauz A, Chaudhry A, Kirson ED, Weinberg U, Palti Y. Mitotic Spindle Disruption by Alternating Electric Fields Leads to Improper Chromosome Segregation and Mitotic Catastrophe in Cancer Cells. Sci Rep. 2015 Dec 11;5:18046. doi: 10.1038/srep18046. PMID 26658786
- [Background] Stupp R, Taillibert S, Kanner AA, Kesari S, Steinberg DM, Toms SA, Taylor LP, Lieberman F, Silvani A, Fink KL, Barnett GH, Zhu JJ, Henson JW, Engelhard HH, Chen TC, Tran DD, Sroubek J, Tran ND, Hottinger AF, Landolfi J, Desai R, Caroli M, Kew Y, Honnorat J, Idbaih A, Kirson ED, Weinberg U, Palti Y, Hegi ME, Ram Z. Maintenance Therapy With Tumor-Treating Fields Plus Temozolomide vs Temozolomide Alone for Glioblastoma: A Randomized Clinical Trial. JAMA. 2015 Dec 15;314(23):2535-43. doi: 10.1001/jama.2015.16669. PMID 26670971
- [Background] Stupp R, Taillibert S, Kanner A, Read W, Steinberg D, Lhermitte B, Toms S, Idbaih A, Ahluwalia MS, Fink K, Di Meco F, Lieberman F, Zhu JJ, Stragliotto G, Tran D, Brem S, Hottinger A, Kirson ED, Lavy-Shahaf G, Weinberg U, Kim CY, Paek SH, Nicholas G, Bruna J, Hirte H, Weller M, Palti Y, Hegi ME, Ram Z. Effect of Tumor-Treating Fields Plus Maintenance Temozolomide vs Maintenance Temozolomide Alone on Survival in Patients With Glioblastoma: A Randomized Clinical Trial. JAMA. 2017 Dec 19;318(23):2306-2316. doi: 10.1001/jama.2017.18718. PMID 29260225